CLINICAL TRIAL: NCT03124680
Title: Opioid Free Anesthesia and Continuous Post-operative Pulse Oximetry Monitoring in the Obese Patient: How About Another Approach?
Brief Title: Opioid Free Anesthesia and Continuous Post-operative Pulse Oximetry Monitoring in the Obese Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Sarah Saxena, Dr, Université Libre de Bruxelles
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OFA
Record Dates: First submitted 2017-03-31; First posted 2017-04-24 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- opioid free group (Active Comparator): Opioid free group using dexmedetomidine, ketamine, lidocaine, MgSO4
  Interventions: Combination Product: Opioid free
- Opioid group (Placebo Comparator): Opioid group using sufentanil, lidocaine, clonidine
  Interventions: Combination Product: opioid group

INTERVENTIONS:
Combination Product: Opioid free — Peroperative opioid free anesthesia will be obtained via a combination of dexmedetomidine, ketamine, lidocaine and magnesium sulfate
  Other Names: study group
  Arms: opioid free group
Combination Product: opioid group — Opioid anesthesia will follow the current standard approach of our hospital.
  Other Names: control group
  Arms: Opioid group

SUMMARY:
Anaesthesia has three major components, analgesia, muscle relaxation and hypnosis.

For a long time, opioids have been covering the analgesia function. (1) When using opioids, an analgesic effect is obtained per-operatively, however, not without side-effects. Post-operative complications such as: respiratory depression, post-operative nausea and vomiting, pruritus, acute opioid tolerance and hyperalgesia, difficulty voiding and ileus, are well known.

Opioid usage is an important risk factor of postoperative desaturation. Postoperative desaturation can lead to severe hypoxemia and even tissue hypoxia, followed by obvious cardiologic and neurological complications.

Thus, in patients at risk, such as the obese patient, experts suggest reducing opioid usage.

Non-opiate protocols implemented on the obese patient have been published. Non-opiate protocols have been established using a combination of ketamine, lidocaine and an alpha-2 agonist.

The main purpose of this pilot study is to evaluate whether patients undergoing an opioid free anaesthesia regime experience less desaturation episodes during the first 24 h post-bariatric surgery than patients having received an opioid anaesthesia regime.

DETAILED DESCRIPTION:
Anaesthesia has three major components, analgesia, muscle relaxation and hypnosis.

For a long time, opioids have been covering the analgesia function. When using opioids, an analgesic effect is obtained per-operatively, however, not without side-effects. Post-operative complications such as: respiratory depression, post-operative nausea and vomiting, pruritus, acute opioid tolerance and hyperalgesia, difficulty voiding and ileus, are well known. These complications may lead to a prolonged hospital stay.

Opioid usage is an important risk factor of postoperative desaturation. Postoperative desaturation can lead to severe hypoxemia and even tissue hypoxia, followed by obvious cardiologic and neurological complications.

Thus, in patients at risk, such as the obese patient, experts suggest reducing opioid usage.

Authors have indeed published non-opiate protocols implemented on the obese patient.

Non-opiate protocols have been established using a combination of ketamine, lidocaine and an alpha-2 agonist.

The main purpose of this pilot study is to evaluate whether patients undergoing an opioid free anaesthesia regime experience less desaturation episodes during the first 24 h post-bariatric surgery than patients having received an opioid anaesthesia regime.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a gastric by-pass surgery will be screened.
* Patients with an ASA physical status of I-II-III (BMI >30) will be included.
* Knowledge of either French, English or Dutch will be required in order to be enrolled in this study.

Exclusion Criteria:

* allergy or contraindications to one of the study drugs
* renal failure
* hepatic failure
* hyperthyroidism
* AV block 2 or 3
* severe bradycardia
* left ventricular failure
* unstable blood pressure
* severe respiratory disease
* epilepsy
* psychiatric disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
desaturation episode evaluation | first 24 hours postoperative
  The primary outcome of this study is to evaluate desaturation episodes during the first 24 h post-bariatric surgery in patients having received an opioid or an opioid free anaesthesia.
  Desaturation is defined as a decrease of oxygen desaturation equal to or exceeding 4% of the baseline value. ODI (oxygen desaturation index), the total number of desaturation events divided by the total time of monitoring in hours, will be calculated to evaluate this outcome in both groups.
  In case of desaturation lasting longer than 10 seconds, oxygen (via nasal canula) will be administered as per post-anaesthesia care unit protocol.
  SP02 will be measured for 24 hours through non-invasive monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided